CLINICAL TRIAL: NCT04233749
Title: The Efficacy of Tranexamic Acid in the Treatment of Lichen Planus Pigmentosus and Erythema Dyschromicum Perstans
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Henry W. Lim, Principal Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15107
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lichen Planus Pigmentosus; Erythema Dyschromicum Perstans; Ashy Dermatosis of Ramirez
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: This a proof-of-concept study. Five subjects will be enrolled and all five will receive tranexamic acid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All five subjects will receive tranexamic acid tablets, 325mg twice daily for six months.
  Interventions: Drug: Tranexamic acid tablets

INTERVENTIONS:
Drug: Tranexamic acid tablets — 325mg of tranexamic acid twice daily for six months
  Other Names: Lysteda, Cyklokapron

SUMMARY:
There are currently no effective treatments for lichen planus pigmentosus (LPP) and erythema dyschromicum perstans (EDP). Tranexamic acid, which may downregulate pigmentation through a reduction in plasmin, has been shown to decrease pigmentation in patients with melasma, another pigmentary disorder. Given that LPP, EDP, and melasma are all disorders of pigmentation with dermal involvement, it is possible that tranexamic acid can also reduce pigmentation in LPP and EDP as well.

DETAILED DESCRIPTION:
Lichen planus pigmentosus (LPP) and erythema dyschromicum perstans (EDP) (also known as ashy dermatosis (AD)) are two conditions on the spectrum of dermal pigmentary disorders. LPP typically affects skin phototypes III-V and has involvement of sun exposed areas or intertriginous areas. It presents as irregularly shaped or oval grey-brown macules and patches that are typically asymptomatic, but can have mild pruritus and burning. EDP, on the other hand, presents as grey-brown macules and patches in sun-protected sites and may have an early inflammatory phase with an erythematous border. It is typically asymptomatic, but can also be mildly pruritic. There is significant histologic overlap between the two conditions including basal cell degeneration, a mild perivascular or band-like infiltrate in the upper dermis, and dermal melanophages.

Multiple treatments for these conditions, including topical corticosteroids, topical calcineurin inhibitors, topical retinoids, chemical peels, minocycline, dapsone, hydroxychloroquine, isotretinoin, griseofulvin, and systemic steroids have been reported in the literature. However, none of these have been effective consistently.

Tranexamic acid (TA) is a synthetic analog of lysine, and serves as a fibrinolytic agent by binding lysine sites on fibrinogen. Commonly used in surgery to prevent bleeding, it has recently been used in dermatology for the treatment of melasma. Melasma is a pigmentary disorder characterized by hyperpigmented patches in sun-exposed areas, often in response to hormones, sunlight, and other factors. The proposed mechanism of action of tranexamic acid in decreasing pigmentation in this condition is that it decreases inflammation by decreasing dermal angiogenesis and inhibits UV induced plasmin activity in keratinocytes. Plasmin activity can increase melanogenic factors, leading to increased pigmentation. In a study by Lee et al., when administered orally at a dose of 250mg twice daily over approximately 4 months, 89.7 % of patients had documented improvement in pigmentation. Of those who improved, the median lightening was approximately 50%, which is significant. Other studies have also shown promising results.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 18 and older
* Subject with a diagnosis of LPP, EDP, or AD
* Subject able to understand requirements of the study and risks involved
* Subject able to sign a consent form
* Subject to have discontinued all topical or oral medications, with the exception of sunscreen, used to treat pigmentary abnormalities one month prior to treatment

Exclusion Criteria:

* Personal history of clotting disorder or thromboembolic disease (deep vein thrombosis (DVT), stroke, etc)
* Active malignancy, excluding non-melanoma skin cancer
* Moderate to severe renal impairment
* History of migraine with aura
* Current anticoagulant therapy
* Current use of hormonal contraception or hormone replacement therapy in the last 30 days
* A woman who is lactating, pregnant, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pigmentation using Colorimetry | 11 visits over 270 days
  Determine if there is a reduction in pigmentation in patients with LPP or EDP after administration of tranexamic acid using colorimetry.
Change in Pigmentation using Diffuse Reflectance Spectroscopy | 11 visits over 270 days
  Determine if there is a reduction in pigmentation in patients with LPP or EDP after administration of tranexamic acid using diffuse reflectance spectroscopy.

SECONDARY OUTCOMES:
Change in Erythema using Colorimetry | 11 visits over 270 days
  Determine if there is a reduction in erythema in patients with LPP or EDP after administration of tranexamic acid using colorimetry.
Change in Erythema using Diffuse Reflectance Spectroscopy | 11 visits over 270 days
  Determine if there is a reduction in erythema in patients with LPP or EDP after administration of tranexamic acid using diffuse reflectance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Henry W Lim, MD, Principal Investigator — Henry Ford HS
Locations (1):
- New Center One, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bala HR, Lee S, Wong C, Pandya AG, Rodrigues M. Oral Tranexamic Acid for the Treatment of Melasma: A Review. Dermatol Surg. 2018 Jun;44(6):814-825. doi: 10.1097/DSS.0000000000001518. PMID 29677015
- [Background] Ghosh A, Coondoo A. Lichen Planus Pigmentosus: The Controversial Consensus. Indian J Dermatol. 2016 Sep-Oct;61(5):482-6. doi: 10.4103/0019-5154.190108. PMID 27688435
- [Background] Kanwar AJ, Dogra S, Handa S, Parsad D, Radotra BD. A study of 124 Indian patients with lichen planus pigmentosus. Clin Exp Dermatol. 2003 Sep;28(5):481-5. doi: 10.1046/j.1365-2230.2003.01367.x. PMID 12950331
- [Background] Kim SJ, Park JY, Shibata T, Fujiwara R, Kang HY. Efficacy and possible mechanisms of topical tranexamic acid in melasma. Clin Exp Dermatol. 2016 Jul;41(5):480-5. doi: 10.1111/ced.12835. Epub 2016 May 2. PMID 27135282
- [Background] Lee HC, Thng TG, Goh CL. Oral tranexamic acid (TA) in the treatment of melasma: A retrospective analysis. J Am Acad Dermatol. 2016 Aug;75(2):385-92. doi: 10.1016/j.jaad.2016.03.001. Epub 2016 May 17. PMID 27206758
- [Background] Molinar VE, Taylor SC, Pandya AG. What's new in objective assessment and treatment of facial hyperpigmentation? Dermatol Clin. 2014 Apr;32(2):123-35. doi: 10.1016/j.det.2013.12.008. PMID 24679999